CLINICAL TRIAL: NCT05293418
Title: Retrospective Single-center Cohort Study to Evaluate the Incidence of Colonization by Multidrug-resistant Organisms in Mechanically Ventilated Patients With Severe COVID-19 Admitted to a Large Intensive Care Unit in Milan, Italy
Brief Title: Incidence of Colonization by Multidrug-resistant Organisms in Mechanically Ventilated Patients With Severe COVID-19
Acronym: MDR_in_Fiera
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 701_2021
Record Dates: First submitted 2022-03-22; First posted 2022-03-24 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Bacterial Infections; Colonization, Asymptomatic
Keywords: COVID-19; mechanical ventilation; multidrug resistance; MDR colonization
MeSH Terms: conditions — COVID-19; Bacterial Infections; Asymptomatic Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU mechanically ventilated COVID-19 patients: Patients admitted to Milano Fiera ICU for COVID-19 requiring mechanical ventilation from October 2020 through May 2021
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection from medical records and the microbiological surveillance system of the enrolled patients

SUMMARY:
Retrospective single-center cohort study to evaluate the incidence of colonization by multidrug-resistant organisms (MDRO) in mechanically ventilated patients admitted to a large intensive care unit (ICU) for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection during the second wave of COVID-19 pandemic (October 2020-May 2021) in Lombardy, Italy. As secondary outcomes, the study evaluates the overall incidence of infections during the ICU stay and assesses the risk factors associated to bacterial superinfection and MDRO colonization.

DETAILED DESCRIPTION:
Bacterial superinfection represents a major treat for patients admitted to intensive care unit (ICU), severely impacting clinical outcome and length of hospital stay. Several studies showed that previous multidrug-resistant organisms (MDRO) colonization is a major risk factor for subsequent infection. The coronavirus disease 2019 (COVID-19) pandemic caused an unprecedented rate of ICU admissions and drastically changed the ICU care itself, in terms of infection control measures and therapeutic usage of immunomodulating drugs. Depending on the study, incidence of bacterial infections acquired in COVID-19 ICUs ranges from 12% to 50%. In a retrospective, multicenter study conducted in 8 Italian ICUs during the first wave of the pandemic (March 2020-May 2020), 46% of the patients developed a bacterial superinfection. Notably, 35% of these infections were caused by MDRO. To date there is still scarce evidence on the incidence of colonization by MDRO in patients admitted to COVID-19 ICUs, and little data has been collected on risk factors associated with MDRO colonization. Based on case series analysis, MDRO colonization has been associated with presence of invasive devices, prolonged ICU stay and use of corticosteroids and antibiotics.

The Milano Fiera ICU was a large, modular, COVID-19 ICU built in Milan, Italy, in March 2020 to face the impact of the pandemic. It was composed of distinct units (modules) to accommodate up to 100 patients with severe SARS-CoV-2 infection requiring mechanical ventilation. Since October 2020, over 400 mechanically ventilated COVID-19 patients were admitted to Milano Fiera ICU. Despite each module was managed by staff coming from different hospitals in the Milan area, microbiological surveillance was standardized, and all modules referred to the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico of Milan for laboratory analysis and infectious disease specialist consultation.

The present retrospective single-center cohort study aims to evaluate the incidence of colonization by MDRO in patients admitted to the Milano Fiera ICU during the second wave of COVID-19 pandemic (October 2020-May 2021). Furthermore, the study will evaluate the overall incidence of infections during the ICU stay and analyze the risk factors associated with bacterial superinfection and with MDRO colonization.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19-related respiratory failure
* Mechanical ventilation at least 48 hours

Exclusion Criteria:

* Age < 18 years
* ICU stay < 48 hours

Concurrent participation in other clinical trials is not a criterion for exclusion from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated COVID-19 patients admitted to Milano Fiera ICU from October 2020 through May 2021
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of MDRO colonization | 1000 patient days
  Crude incidence rate of MDRO colonization will be calculated globally and subdivided by hospital of provenance, module of hospitalization and microbiological criteria.

SECONDARY OUTCOMES:
Incidence of bacterial infections | 1000 patient days
  Crude incidence rate of bacterial infections (both MDR and antibiotic-susceptible bacteria) will be calculated globally and subdivided by hospital of provenance, module of hospitalization and microbiological criteria.
risk factors for MDRO colonization and bacterial infections | 1000 patient days
  Cumulative incidence rate of MDRO colonization and bacterial infections, obtained from multivariable models that consider the competitive effect of death on colonization (main event). The model will provide for each analyzed predictor (i.e., patient conditions at enrollment, previous exposition to corticosteroid and/or antibiotic therapy, biochemical indexes) the corresponding sub-hazard ratio

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaola Monti, MD, Principal Investigator — Intensive Care Unit, ASST Grande Ospedale Metropolitano Niguarda - Milano (Italy); Andrea Gori, MD, Principal Investigator — Infectious Diseases Unit, IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation - Milano (Italy)
Locations (1):
- IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be shared upon written request to the study director

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Onder G, Rezza G, Brusaferro S. Case-Fatality Rate and Characteristics of Patients Dying in Relation to COVID-19 in Italy. JAMA. 2020 May 12;323(18):1775-1776. doi: 10.1001/jama.2020.4683. No abstract available. PMID 32203977
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Grasselli G, Scaravilli V, Mangioni D, Scudeller L, Alagna L, Bartoletti M, Bellani G, Biagioni E, Bonfanti P, Bottino N, Coloretti I, Cutuli SL, De Pascale G, Ferlicca D, Fior G, Forastieri A, Franzetti M, Greco M, Guzzardella A, Linguadoca S, Meschiari M, Messina A, Monti G, Morelli P, Muscatello A, Redaelli S, Stefanini F, Tonetti T, Antonelli M, Cecconi M, Foti G, Fumagalli R, Girardis M, Ranieri M, Viale P, Raviglione M, Pesenti A, Gori A, Bandera A. Hospital-Acquired Infections in Critically Ill Patients With COVID-19. Chest. 2021 Aug;160(2):454-465. doi: 10.1016/j.chest.2021.04.002. Epub 2021 Apr 20. PMID 33857475
- [Background] Rouze A, Martin-Loeches I, Povoa P, Makris D, Artigas A, Bouchereau M, Lambiotte F, Metzelard M, Cuchet P, Boulle Geronimi C, Labruyere M, Tamion F, Nyunga M, Luyt CE, Labreuche J, Pouly O, Bardin J, Saade A, Asfar P, Baudel JL, Beurton A, Garot D, Ioannidou I, Kreitmann L, Llitjos JF, Magira E, Megarbane B, Meguerditchian D, Moglia E, Mekontso-Dessap A, Reignier J, Turpin M, Pierre A, Plantefeve G, Vinsonneau C, Floch PE, Weiss N, Ceccato A, Torres A, Duhamel A, Nseir S; coVAPid study Group. Relationship between SARS-CoV-2 infection and the incidence of ventilator-associated lower respiratory tract infections: a European multicenter cohort study. Intensive Care Med. 2021 Feb;47(2):188-198. doi: 10.1007/s00134-020-06323-9. Epub 2021 Jan 3. PMID 33388794
- [Background] Bogossian EG, Taccone FS, Izzi A, Yin N, Garufi A, Hublet S, Njimi H, Ego A, Gorham J, Byl B, Brasseur A, Hites M, Vincent JL, Creteur J, Grimaldi D. The Acquisition of Multidrug-Resistant Bacteria in Patients Admitted to COVID-19 Intensive Care Units: A Monocentric Retrospective Case Control Study. Microorganisms. 2020 Nov 19;8(11):1821. doi: 10.3390/microorganisms8111821. PMID 33227956
- [Background] Baiou A, Elbuzidi AA, Bakdach D, Zaqout A, Alarbi KM, Bintaher AA, Ali MMB, Elarabi AM, Ali GAM, Daghfal J, Almaslamani MA, Ibrahim ASS, Alkhal A, Omrani AS. Clinical characteristics and risk factors for the isolation of multi-drug-resistant Gram-negative bacteria from critically ill patients with COVID-19. J Hosp Infect. 2021 Apr;110:165-171. doi: 10.1016/j.jhin.2021.01.027. Epub 2021 Feb 6. PMID 33561503
- [Background] Karruli A, Boccia F, Gagliardi M, Patauner F, Ursi MP, Sommese P, De Rosa R, Murino P, Ruocco G, Corcione A, Andini R, Zampino R, Durante-Mangoni E. Multidrug-Resistant Infections and Outcome of Critically Ill Patients with Coronavirus Disease 2019: A Single Center Experience. Microb Drug Resist. 2021 Sep;27(9):1167-1175. doi: 10.1089/mdr.2020.0489. Epub 2021 Feb 17. PMID 33600262
- [Background] Patel A, Emerick M, Cabunoc MK, Williams MH, Preas MA, Schrank G, Rabinowitz R, Luethy P, Johnson JK, Leekha S. Rapid Spread and Control of Multidrug-Resistant Gram-Negative Bacteria in COVID-19 Patient Care Units. Emerg Infect Dis. 2021 Apr;27(4):1234-1237. doi: 10.3201/eid2704.204036. Epub 2021 Feb 10. PMID 33565961
- [Background] Austin PC, Fine JP. Practical recommendations for reporting Fine-Gray model analyses for competing risk data. Stat Med. 2017 Nov 30;36(27):4391-4400. doi: 10.1002/sim.7501. Epub 2017 Sep 15. PMID 28913837
- [Background] Amorim LD, Cai J. Modelling recurrent events: a tutorial for analysis in epidemiology. Int J Epidemiol. 2015 Feb;44(1):324-33. doi: 10.1093/ije/dyu222. Epub 2014 Dec 9. PMID 25501468